CLINICAL TRIAL: NCT03283696
Title: A Phase 1b Study of Olaratumab, Doxorubicin and Ifosfamide in the Treatment of Patients With Advanced or Metastatic Soft Tissue Sarcoma
Brief Title: A Study of Olaratumab (LY3012207), Doxorubicin, and Ifosfamide in Participants With Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16430; I5B-MC-JGDR (Other: Eli Lilly and Company); 2016-004287-19 (EudraCT Number)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Doxorubicin; Ifosfamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaratumab + Doxorubicin + Ifosfamide + Mesna (Experimental): Olaratumab 15 milligrams per kilogram (mg/kg) on Days 1 and 8 of a 21-day cycle, in combination with doxorubicin and ifosfamide was administered. When the safety of the 15-mg/kg dose of olaratumab was established, a 20-mg/kg loading dose cycle of olaratumab on Days 1 and 8 of a 21-day cycle in Cycle 1 only, followed by 15 mg/kg on Days 1 and 8 of subsequent cycles in combination with doxorubicin and ifosfamide plus mesna, was administered.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin; Drug: Ifosfamide; Drug: Mesna

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207
Drug: Doxorubicin — Administered IV
Drug: Ifosfamide — Administered IV
Drug: Mesna — Administered per standard of care

SUMMARY:
The purpose of this study is to evaluate the safety of ifosfamide when added to the combination regimen of olaratumab and doxorubicin in participants with advanced or metastatic soft tissue sarcoma (STS).

ELIGIBILITY:
Inclusion Criteria:

* Have a histological diagnosis of advanced STS (by local pathology review), for which treatment with doxorubicin, ifosfamide and mesna is deemed appropriate by the investigator.
* Have measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Have adequate hematologic, organ and coagulation function within 2 weeks (14 days) prior to enrollment.
* Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group scale.
* Have received no prior lines of systemic therapy and are suitable to receive doxorubicin, ifosfamide and mesna. All previous anticancer treatments must have completed ≥3 weeks (21 days) prior to the first dose of study treatment.
* Have left ventricular ejection fraction (LVEF) ≥50% assessed within 28 days prior to enrollment.
* Have resolution of Adverse Events (AEs), with the exception of alopecia, and of all clinically significant toxic effects of prior locoregional therapy, surgery or radiotherapy to ≤Grade 1, by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0.
* Have sufficient available material from archived formalin-fixed paraffin-embedded tumor tissue for biomarker-related studies. If such tissue is not available, a newly obtained core or excisional biopsy of a tumor lesion must be performed.
* If male, must be sterile or agree to use an effective method of contraception or a highly effective method of contraception during the study and for at least 12 weeks following the last dose of study treatment.
* If female and of child-bearing potential, must:

  1. have a negative serum pregnancy test at the time of enrollment,
  2. have a negative urine pregnancy test within 24 hours prior to the first dose of study treatment, and
  3. agree to use a highly effective method of contraception during the study and for 3 months following the last dose of study treatment.
* Have a life expectancy of at least 3 months, in the opinion of the investigator.

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated within the past 30 days in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed.
* Have previously completed or withdrawn from any study investigating olaratumab.
* Have received prior treatment with olaratumab, doxorubicin, or ifosfamide, or have participated in other trials investigating olaratumab.
* Have received prior radiotherapy of the mediastinal/pericardial area or whole pelvis radiation.
* Have known urinary outflow obstruction, or inflammation of the urinary bladder (cystitis).
* Are diagnosed with gastrointestinal stromal tumor or Kaposi sarcoma.
* Have active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of enrollment. Participants with a history of CNS metastasis (previously treated with curative intent [for example, stereotactic radiation or surgery]) that has not progressed on follow-up imaging, have been asymptomatic for at least 60 days, and are not receiving systemic corticosteroids and/or anticonvulsants are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before enrollment to rule out brain metastasis.
* Have a history of another primary malignancy, with the exception of:

  1. curatively treated non-melanomatous skin cancer
  2. curatively treated cervical carcinoma in situ
* Have an active fungal, bacterial and/or known viral infection including human immunodeficiency virus or viral (A, B, or C) hepatitis (screening is not required).
* Have Grade 3 or 4 peripheral neuropathy per NCI-CTCAE Version 4.0.
* Have a serious cardiac condition.
* Have a resting heart rate of >100 beats per minute (bpm).
* Have a Fridericia's QT corrected interval (QTcF) interval of >450 milliseconds (msec) for males and >470 msec for females on screening electrocardiogram (ECG) utilizing Fridericia's correction.
* Have uncontrolled intercurrent illness including, but not limited to, an ongoing/active infection requiring parenteral antibiotics.
* Have a psychiatric illness/social situation that would limit compliance with study requirements.
* Have electively planned or will require major surgery during the course of the study.
* Are females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (2):
  - University of Miami School of Medicine, Miami, Florida
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (2):
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - HELIOS Klinikum Berlin-Buch, Berlin
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan, Lombardy
  - Università degli Studi di Catania - Azienda Policlinico, Catania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Olaratumab (LY3012207), Doxorubicin, and Ifosfamide in Participants With Advanced or Metastatic Soft Tissue Sarcoma — https://www.lillytrialguide.com/en-US/studies/soft-tissue-sarcoma/JGDR#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause, participants with progressive disease.
Groups:
- Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide: Participants received olaratumab 15 milligrams per kilogram (mg/kg) on days 1, 8 plus doxorubicin 25 milligrams per meter square (mg/m^2) on days 1, 2, 3 plus ifosfamide 2.5 gram per meter square (g/m^2) per day on days 1, 2, 3, 4 plus mesna dose ≥ 60% of ifosfamide dose on days 1, 2, 3 of a 21-day cycle for a maximum of 6 cycles, or until a discontinuation criterion was met. All treatments were administered intravenously.
- Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide: Participants received olaratumab 20 mg/kg loading dose on days 1, 8 of cycle 1. From cycle 2, they received olaratumab 15 mg/kg on days 1, 8 plus doxorubicin 25 mg/m^2 on days 1, 2, 3 plus ifosfamide 2.5 g/m^2 per day on days 1, 2, 3, 4 plus mesna dose ≥60% of ifosfamide dose on days 1, 2, 3 of a 21-day cycle for a maximum of 6 cycles, or until a discontinuation criterion was met. All treatments were administered intravenously.
Period: Overall Study
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Started | 16 | 8
Received at Least 1 Dose of Study Drug | 16 | 8
Completed | 9 | 2
Not Completed | 7 | 6
Not completed — Physician Decision | 5 | 6
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide: Participants received olaratumab 15 mg/kg on days 1, 8 plus doxorubicin 25 mg/m^2 on days 1, 2, 3 plus ifosfamide 2.5 g/m^2 per day on days 1, 2, 3, 4 plus mesna dose ≥ 60% of ifosfamide dose on days 1, 2, 3 of a 21-day cycle for a maximum of 6 cycles, or until a discontinuation criterion was met. All treatments were administered intravenously.
- Total: Total of all reporting groups
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.1) | 49.8 (11.1) | 45.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 8 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
  Italy | 3 | 0 | 3
  Germany | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Olaratumab Dose Limiting Toxicities (DLTs)
Description: A Dose Limiting Toxicity is defined as an Adverse Event (AE) that is likely related to the study medication or combination, and fulfills any one of the following criteria, graded according to the NCI-CTCAE Version 4.0:
  1. Grade 3 or 4 febrile neutropenia, or sepsis., or
  2. Grade 4 neutropenia lasting 7 days or longer.
  3. Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia complicated by hemorrhage.
  4. Nonhematologic Grade ≥3 toxicity, except for toxicities (such as nausea, vomiting, transient electrolyte abnormalities, or diarrhoea) that can be controlled with optimal medical management within 48 hours or clinically non-significant laboratory abnormalities.
Time Frame: Cycle 1 (Up To 24 days)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Participants | 4 | 4

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Olaratumab
Description: PK: Cmax of olaratumab.
Time Frame: Cycle 1 - Day 1 (predose, end of infusion, 2 hours post olaratumab (olara), 6 hours post olara, 24 hours post olara, 72 hours post olara), Day 8 (predose, end of infusion, 2 hours post-olara, 6 hours post olara, 48 hours post olara, 168 hours post olara)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
micrograms per milliliter (μg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 14 | 8
  Cycle 1 Day 1 | 408 (25) | 508 (27)
  Cycle 1 Day 8: number analyzed (Participants) | 12 | 6
  Cycle 1 Day 8 | 452 (28) | 671 (24)

3. Secondary Outcome: PK: Maximum Serum Concentration (Cmax,ss) of Olaratumab at Steady-state
Description: PK: Cmax of olaratumab at steady-state.
Time Frame: Cycle 3 - Day 1 (predose, end of infusion, 2 hours post olara, 5 hours post olara, 24 hours post olara, 72 hours post olara), Day 8 (predose, end of infusion, 2 hours post-olara, 5 hours post olara, 48 hours post olara, 168 hours post olara)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
micrograms per milliliter (μg/mL)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 7
  Cycle 3 Day 1 | 533 (22) | 494 (9)
  Cycle 3 Day 8: number analyzed (Participants) | 14 | 5
  Cycle 3 Day 8 | 523 (18) | 545 (13)

4. Secondary Outcome: PK: Trough Serum Concentration (Cmin)
Description: PK: Cmin of olaratumab.
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
micrograms per milliliter (μg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 11 | 6
  Cycle 1 Day 1 | 87.3 (40) | 140 (45)
  Cycle 1 Day 8: number analyzed (Participants) | 16 | 6
  Cycle 1 Day 8 | 46.7 (105) | 53.3 (143)

5. Secondary Outcome: PK: Trough Serum Concentration (Cmin,ss) of Olaratumab at Steady-state
Description: PK: Cmin of olaratumab at steady-state.
Time Frame: as for outcome 3
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
micrograms per milliliter (μg/mL)
  Cycle 3 Day 1: number analyzed (Participants) | 14 | 6
  Cycle 3 Day 1 | 154 (26) | 177 (17)
  Cycle 3 Day 8: number analyzed (Participants) | 14 | 7
  Cycle 3 Day 8 | 126 (35) | 115 (32)

6. Secondary Outcome: Number of Participants With Anti-Olaratumab Antibodies
Description: Participants with treatment-emergent anti-drug antibody (TE ADA) positive were 1) a participant with a 4-fold (2 dilutions) increase over a positive baseline antibody titer; or 2) for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Baseline through Follow-up (Up To 21 Months)
Population: All participants with an evaluable baseline and at least 1 post-baseline data for Anti-Olaratumab Antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 15 | 8
Participants | 0 | 1

7. Secondary Outcome: Objective Response Rate (ORR): Number of Participants Who Achieve Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR)
Description: Objective response rate is the best overall tumor response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions.
Time Frame: Baseline up to Short-Term Follow-Up Period (Up To 21 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Participants | 6 | 1

8. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival time was measured from randomization until the date of objective progression as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), or death from any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Participants who have neither progressed nor died were censored at the day of their last radiographic tumor assessment, if available, or date of randomization if no post-baseline radiographic assessment is available.
Time Frame: Baseline to Objective Disease Progression or Death Due to Any Cause (Up To 21 Months)
Population: All participants who received at least one dose of study drug. Number of participants censored were Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide = 8 and Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide = 6.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Months | 9.53 [4.07 to 14.29] | 6.93 [1.28 to 6.93]

9. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the date measurement criteria for CR or PR (whichever is first recorded) are first met until the first date that disease is recurrent or objective progression is observed, per RECIST 1.1, or the date of death from any cause in the absence of objectively determined disease progression or recurrence. Participants known to be alive and without disease progression will be censored at the time of the last adequate tumor assessment.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Objective Disease Progression or Death Due to Any Cause (Up To 21 Months)
Population: All participants who received at least one dose of study drug. Number of participants censored were Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide = 4 and Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide = 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Months | 8.25 [8.15 to 8.34] | NA [NA to NA] — Values not attained due to high censoring rate.

10. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD)
Description: Disease control rate (DCR) is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline until Disease Progression or Death Due to Any Cause (Up To 21 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Percentage of participants | 81.3 | 87.5

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. For each participant who is not known to have died as of the data-inclusion cut-off date for a particular analysis, overall survival duration was censored for that analysis at the date of last prior contact.
Time Frame: Baseline to Date of Death Due to Any Cause (Up To 21 Months)
Population: All participants who received at least one dose of study drug. Number of participants censored were Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide = 9 and Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide = 6.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
Number analyzed (Participants) | 16 | 8
Months | 16.72 [8.38 to NA] — Values not attained due to high censoring rate. | NA [1.28 to NA] — Values not attained due to high censoring rate.

ADVERSE EVENTS:
Time Frame: Up To 2 years
Description: All participants who received at least one dose of study drug. There are gender specific adverse events, occurring only in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide
All-Cause Mortality (participants affected / at risk) | 7/16 | 2/8
Serious Adverse Events (participants affected / at risk) | 9/16 | 7/8
Other Adverse Events (participants affected / at risk) | 16/16 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide (N=16) | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (8) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 2 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olaratumab 15 mg/kg + Doxorubicin + Ifosfamide (N=16) | Olaratumab 20 mg/kg + Doxorubicin + Ifosfamide (N=8)
Anaemia (Blood and lymphatic system disorders) | 11 (63) | 8 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 3 (6)
Lymphopenia (Blood and lymphatic system disorders) | 3 (8) | 2 (7)
Neutropenia (Blood and lymphatic system disorders) | 9 (26) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (20) | 3 (13)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Dry eye (Eye disorders) | 2 (3) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (26) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (39) | 6 (16)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 2 (6) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (15) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (12) | 3 (4)
Asthenia (General disorders) | 4 (8) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 12 (22) | 6 (16)
Mucosal inflammation (General disorders) | 5 (5) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1/7 (3) | 0/3 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1/9 (1) | 0/5 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (9) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram st segment depression (Investigations) | 1 (1) | 0 (0)
Electrocardiogram t wave amplitude decreased (Investigations) | 1 (1) | 0 (0)
Hormone level abnormal (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 1 (7)
Platelet count decreased (Investigations) | 1 (2) | 2 (15)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (5) | 2 (10)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 2 (7) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (9) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (6) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (3)
Paraparesis (Nervous system disorders) | 1 (2) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1/9 (1) | 0/5 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT03283696/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03283696/SAP_001.pdf